CLINICAL TRIAL: NCT03281863
Title: Clinical Audit on the Managment of Rheumatic Fever in Assiut University Children Hospital
Brief Title: Clinical Audit on the Managment in Assiut University Children Hospital
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Patricia reda hanna, Resident doctor, Assiut University
Other Study IDs: AssiutU71516
Record Dates: First submitted 2017-08-29; First posted 2017-09-13 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Rheumatic Fever
MeSH Terms: conditions — Rheumatic Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: C reactive protein, anti streptolysin o antibody test ,erythrocyte sedimentation rate — Throat culture to detect the causative organism
  Other Names: Throat culture

SUMMARY:
clinical audit on the Managment of rheumatic fever in assiut university children hospital.

DETAILED DESCRIPTION:
Acute rheumatic fever,an auto immune response to Group A streptococcus infection of the upper respiratory tract,may result in carditis.when the inflammation leads to permenant damage of the valves the individual has rheumatic heart disease.

Recurrences of rheumatic fever are likely in the absence of preventive measures and may cause further cardiac valve and muscle damage,leading to heart failure,stroke and premature death.bacterial endocarditis is also a complication.

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed diagnosis of rheumatic fever based on laboratory investigations.

Exclusion Criteria:

* No

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Clinical audit on the managment of rheumatic fever in assiut university children hospital
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
laboratory investigations (ASOt , ESR . CRP) | One year from October 2017 to september 2018
  laboratory investigations that measure the inflammation process will be used and the target that the ASOt not increase 1/400

SECONDARY OUTCOMES:
clinical measures | One year from October 2017 to september 2018
  improvement of arthritis if found

CONTACTS AND LOCATIONS:
Locations (1):
- Egypt, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No